CLINICAL TRIAL: NCT03002090
Title: Defining the Functional and Metabolic Role of Iron in Aerobic Training and Physical Performance
Brief Title: Defining the Functional Role of Iron in Aerobic Training and Physical Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB #: 1402004495
Record Dates: First submitted 2016-12-14; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Iron Deficiency Without Anemia
Keywords: iron deficiency; anemia; exercise training; aerobic; performance; Chinese medicine; BaZhen KeLi
MeSH Terms: conditions — Iron Deficiencies; Anemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Iron trained (Experimental)
  Interventions: Dietary Supplement: Iron trained
- Iron Untrained (Experimental)
  Interventions: Dietary Supplement: Iron Untrained
- BZKL Trained (Experimental)
  Interventions: Dietary Supplement: BZKL Trained
- BZKL Untrained (Experimental)
  Interventions: Dietary Supplement: BZKL Untrained
- Placebo Trained (Experimental)
  Interventions: Dietary Supplement: Placebo Trained
- Placebo Untrained (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Untrained

INTERVENTIONS:
Dietary Supplement: Iron trained — 1. Ferrous sulfate: 100 mg/day of FeSO4 dosed in 2 capsules taken individually by mouth with breakfast and dinner. Capsules were made with FeSO4 and dextrose. Analysis has shown that each capsule contains 11mg of elemental iron, which is expected to be absorbed at roughly 33% bioavailability.
  2. Aerobic Training: 25 minutes/day, 5 days/week for 8 weeks working at an intensity between 75-85% of age-predicted maximum heart rate.
  Arms: Iron trained
Dietary Supplement: Iron Untrained — 1. Ferrous sulfate: 100 mg/day of FeSO4 dosed in 2 capsules taken individually by mouth with breakfast and dinner. Capsules were made with FeSO4 and dextrose. Analysis has shown that each capsule contains 11mg of elemental iron, which is expected to be absorbed at roughly 33% bioavailability.
  Arms: Iron Untrained
Dietary Supplement: BZKL Trained — 1. BaZhen KeLi capsules: Traditional Chinese herbal supplement composed of: Radix Paeoniae Alba (White peony root), Rhizoma Atractylodis (Atractylodes), Rhizoma Chuanxiong (Chuanxiong), Radix Angelicae Sinensis (Angelica), Radix Codonopsis Pilosula (Codonopsis), Poria cocos (Poria), licorice, and Rehmannia glutinosa Each pill contained 5g of licorice and 10g of all other ingredients. Dosed in 2 capsules taken individually by mouth with breakfast and dinner. Analysis has shown that each capsule contained 0.5mg of elemental iron.
  2. Aerobic Training: 25 minutes/day, 5 days/week for 8 weeks working at an intensity between 75-85% of age-predicted maximum heart rate.
  Arms: BZKL Trained
Dietary Supplement: BZKL Untrained — 1. BaZhen KeLi capsules: Traditional Chinese herbal supplement composed of: Radix Paeoniae Alba (White peony root), Rhizoma Atractylodis (Atractylodes), Rhizoma Chuanxiong (Chuanxiong), Radix Angelicae Sinensis (Angelica), Radix Codonopsis Pilosula (Codonopsis), Poria cocos (Poria), licorice, and Rehmannia glutinosa Each pill contained 5g of licorice and 10g of all other ingredients. Dosed in 2 capsules taken individually by mouth with breakfast and dinner. Analysis has shown that each capsule contained 0.5mg of elemental iron.
  Arms: BZKL Untrained
Dietary Supplement: Placebo Trained — 1. Aerobic Training: 25 minutes/day, 5 days/week for 8 weeks working at an intensity between 75-85% of age-predicted maximum heart rate.
  Arms: Placebo Trained
Dietary Supplement: Placebo Untrained — No intervention
  Arms: Placebo Untrained

SUMMARY:
Iron deficiency is known to negatively impact physical performance, attention, and time spent doing physical activity. As a result, an iron deficient person must expend more energy to complete the same amount of work as someone who is healthy. Another interesting relationship has been observed between exercise training and iron status in that women who participate in exercise training often have higher rates of iron deficiency than sedentary women. ID is commonly treated using daily iron supplementation. However, it is currently unknown whether participating in regular exercise somehow impacts the effectiveness of iron supplementation. Iron deficient women who participate in exercise programs may potentially benefit less from iron supplementation than those who do not. Another common treatment for the symptoms of iron deficiency is the traditional Chinese herbal treatment, Ba-Zhen-Ke-Li (BZKL). While studies have shown that BZKL impacts expression of some iron-related proteins and increases endurance performance in rats, no studies have examined the efficacy of BZKL in improving iron markers or physical performance in humans. This study will compare the efficacy of BZKL in improving iron status and physical performance with that of ferrous sulfate supplementation. The Cornell research team will achieve these objectives in collaboration with colleagues at Kunming Medical University (KMU) in Kunming, China. A double-blind, randomized, placebo controlled study will be conducted by a Cornell graduate student at KMU. The subjects will be healthy women, age 18-26 years, attending KMU. Blood samples will be collected and analyzed for measures of iron).

Subjects will be randomly assigned to receive 50 mg of ferrous sulfate (10 mg of elemental iron), 6mg of BZKL, or an identical placebo pill twice daily for 8 weeks. Subjects will be further randomly sub-divided to receive aerobic exercise training or no training during the 8-week supplementation period. At weeks 4 and 8, subjects will perform the same series of tests as was performed at baseline. The investigators hypothesize that: 1. the women who train and received iron will have smaller improvements in iron status than those who do not train 2. The women who receive iron and train will have greater improvements in physical performance than those who train and do not receive iron, and 3. The women who receive BZKL will improve their iron status or physical performance more than those who receive placebo.

DETAILED DESCRIPTION:
Background: Despite the overall improvements in malnutrition in the Chinese population, iron deficiency (ID) and iron deficiency anemia (low iron and low hemoglobin, IDA) are still widely prevalent in China. According to recent studies, the prevalence of anemia in Chinese women of childbearing age is 20% and can be as high as 30% in rural areas, with 85% of anemia cases resulting from ID. Diabetes, heart disease, and obesity are also highly prevalent in China - though the Chinese government is taking actions against these epidemics, often via interventions promoting physical activity. Iron deficiency without anemia (IDNA) can impair adult physical performance and lowers time spent doing voluntary physical activities. However, iron supplementation intended to alleviate IDNA may be less effective in those who are physically active, suggesting an intricate, but currently undefined, relationship between iron status, exercise, and physical performance capacity. A combined analysis of iron status, exercise training, and physical performance in Chinese women could illuminate interactions between these factors and their role in diabetes and obesity reduction.

One common treatment for the symptoms of iron deficiency is the traditional Chinese herbal treatment, Ba-Zhen-Ke-Li (BZKL). While studies have shown that BZKL impacts expression of some iron-related proteins and increases endurance performance in rats, no studies have examined the efficacy of BZKL in improving iron markers or physical performance in humans. This study will compare the efficacy of BZKL in improving iron status and physical performance with that of ferrous sulfate supplementation.

Significance and Specific Aims:

The goal of the proposed research is to clarify the relationship between iron status, physical performance, and aerobic exercise training. By conducting an iron intervention study in combination with an exercise training program, the investigators can examine the modifying effect of iron status on the physical performance changes from aerobic exercise training as well as the modifying effect of participation in aerobic exercise in maintenance of iron status. To achieve this goal, a randomized double-blind, placebo controlled trial will be conducted with Chinese collegiate women.

The proposed work will be organized along three specific aims:

Aim I: To determine how changes in iron status, alone or in combination with exercise training, influence physical performance. Hypothesis: Subjects who both improve iron status and receive exercise training will show improvements in physical performance greater than the additive improvements resulting from either treatment alone. This result would suggest iron replete individuals benefit more from exercise training than those who are iron deficient.

Aim II: To determine how aerobic exercise training affects the maintenance of iron homeostasis. Hypothesis: Subjects participating in exercise training will show smaller improvements in iron status from iron supplementation than sedentary subjects who receive the same iron supplementation. This would suggest regular exercise training negatively impacts iron absorption, iron excretion and/or iron homeostasis.

Aim III: To determine whether BZKL can be used as an alternative to iron supplementation for improving iron status or physical performance of iron deficient, non-anemic women. Hypothesis: Those women who receive BZKL will improve in iron status and physical performance measures more than those who receive placebo.

The proposed research in Aims 1 and 2 is important because there is no known explanation for the observed relationships between iron, exercise training, and physical performance in IDNA. This research will allow clarification of the role that iron status plays in modifying the effects of exercise training on physical performance as well as whether participation in exercise impacts effectiveness of iron supplementation in improving iron status.

The long-term significance of this research is that establishing these relationships will further the current understanding of how iron status impacts and is impacted by aerobic exercise and physical performance. This knowledge could lead to improved physical activity interventions, which help reduce chronic diseases like obesity and diabetes in populations with high prevalence of ID, such as the U.S. and China. It will also help to inform iron interventions designed to alleviate ID in physically active populations, such as rural Chinese laborers and women in developed countries who participate in aerobic training to improve fitness.

Research Design and Methods:

Participants will be female subjects between the ages of 18-26 years with low body iron but normal hemoglobin (Hb) levels, (ferritin <20 μg/L and Hb > 120 g/L) who are otherwise healthy.

The study will be a randomized double-blind, placebo controlled trial with a 3x2 design. Power calculations were based on the pilot study performed by the investigators in Shanghai in 2013 and a study by Brownlie et al. Sample size was calculated to require 24 women per group, which was expanded to 29 subjects per group to allow for sample dropout. Subjects will be randomized to receive either 50mg of ferrous sulfate capsule twice a day (20mg elemental iron/day), 6 mg of BaZhen KeLi, or identical placebo capsules for 8 weeks. Half of each supplement group will also be randomly assigned to receive 8 weeks of aerobic exercise training (5 days/week, 25 minutes/day) or no training.

At weeks 0, 4, and 8 subjects will complete the following:

1. Anthropometric measurements (height, weight, skinfold thickness)
2. Physical activity and 4-day dietary intake questionnaires
3. Resting venous blood draw for iron status assessment
4. Exercise testing (VO2max test and energetic efficiency test)

To address Aims 1 and 2, the investigators will compare energetic efficiency, maximum ability to use oxygen, ventilatory threshold, and blood lactate concentrations at baseline, after supplementation (or placebo), and after exercise training (or no training). The 3x2 study design will allow for the determination of whether subjects receiving iron benefit more from exercise training. The investigators will also examine whether participating in exercise training affects iron homeostasis or lowers iron status.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-26
* Must be able to complete exercise on a stationary bicycle
* Clinical diagnosis of iron depletion without severe anemia (sFer< 25µg/L, Hb>110g/L)
* Willing to comply with the 8-week supplementation and if assigned, training program

Exclusion Criteria:

* age less than 18
* severe anemia (Hb<90g/L in blood analyses)
* current pregnancy or pregnancy within the previous year
* recent infectious illness or fever
* current inflammation or chronic inflammatory diseases (AGP > 1.0 g/L in blood analyses)
* hemolytic anemia
* chronic respiratory disease
* musculoskeletal problems
* history of eating disorders
* smoking, BMI < 18 or >24 kg/m2
* consumption of medications that may affect dietary iron intake or absorption or that have anticoagulant properties
* participation in varsity sports team

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Concentration of serum ferritin in µg/L | Change in concentration of the 5 biomarkers from weeks 0 to 8. Change in concentration of the 5 biomarkers from weeks 0 to 4.
  Changes from week 0 to weeks 4 and 8 measured both within and between groups.
Concentration of soluble transferrin receptor in mg/L | Change in concentration of the 5 biomarkers from weeks 0 to 8. Change in concentration of the 5 biomarkers from weeks 0 to 4.
  Changes from week 0 to weeks 4 and 8 measured both within and between groups.
Concentration of hemoglobin g/L | Change in concentration of the 5 biomarkers from weeks 0 to 8. Change in concentration of the 5 biomarkers from weeks 0 to 4.
  Changes from week 0 to weeks 4 and 8 measured both within and between groups.
Concentration of alpha-1-acid glycoprotein in g/L | Change in concentration of the 5 biomarkers from weeks 0 to 8. Change in concentration of the 5 biomarkers from weeks 0 to 4.
  Changes from week 0 to weeks 4 and 8 measured both within and between groups.
Concentration of C-reactive protein in mg/L | Change in concentration of the 5 biomarkers from weeks 0 to 8. Change in concentration of the 5 biomarkers from weeks 0 to 4.
  Changes from week 0 to weeks 4 and 8 measured both within and between groups.

SECONDARY OUTCOMES:
Human performance as assessed by maximal capacity for oxygen uptake (mL/min/kg body weight) | Change from weeks 0 to 8. Change from weeks 0 to 4.
  Changes from week 0 to weeks 4 and 8 measured both within and between groups.
Human performance as assessed by energetic efficiency (in %) | Change from weeks 0 to 8. Change from weeks 0 to 4.
  Changes from week 0 to weeks 4 and 8 measured both within and between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jere Haas, PhD, Principal Investigator — Cornell University
Locations (1):
- Kunming Medical University, Department of Nursing,, Longcheng, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pompano LM, Haas JD. Increasing Iron Status through Dietary Supplementation in Iron-Depleted, Sedentary Women Increases Endurance Performance at Both Near-Maximal and Submaximal Exercise Intensities. J Nutr. 2019 Feb 1;149(2):231-239. doi: 10.1093/jn/nxy271. PMID 30649365
- [Derived] Pompano LM, Haas JD. Efficacy of iron supplementation may be misinterpreted using conventional measures of iron status in iron-depleted, nonanemic women undergoing aerobic exercise training. Am J Clin Nutr. 2017 Dec;106(6):1529-1538. doi: 10.3945/ajcn.117.152777. Epub 2017 Nov 1. PMID 29092885